CLINICAL TRIAL: NCT03212001
Title: TeleHomecaRe InterVention Evaluation (THRIVE) Study
Brief Title: TeleHomecaRe InterVention Evaluation Study
Acronym: THRIVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Dr. Valeria Rac, Associate Program Director, University of Toronto
Other Study IDs: 16-5136
Record Dates: First submitted 2017-03-27; First posted 2017-07-11 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Telehomecare patients (matched cohort study): COPD and HF patients in Telehomecare program (followed up to 18 months)
- Usual-care patients (matched cohort study): COPD and HF patients in 'usual care' (followed up to 18 months)
- Telehomecare patients (observations, interviews and surveys): 1. Observational fieldwork conducted to observe everyday routine activities related to Telehomecare.
  2. In-depth interview conducted for 30-60 min using semi-structured interview guide to assess patient experience with Telehomecare program.
  3. Surveys conducted up to four times using validated survey tools.
- Informal caregiver (observations, interviews and surveys): 1. Observational fieldwork conducted to observe everyday routine activities related to Telehomecare.
  2. In-depth interview conducted for 30-60 min using semi-structured interview guide to assess caregiver experience with Telehomecare program.
  3. Surveys conducted up to four times using validated survey tools.
- Healthcare providers (observations, interviews and surveys): 1. Observational fieldwork conducted to observe everyday routine activities related to Telehomecare.
  2. In-depth interview conducted for 30-60 min using semi-structured interview guide to assess provider experience with Telehomecare program.
- Administrators and Decision Makers (observations, interviews): 1. Observational fieldwork conducted to observe everyday routine activities related to Telehomecare.
  2. In-depth interview conducted for 30-60 min using semi-structured interview guide to assess administrator/decision-maker experience with Telehomecare program.
- Technician (observation, interviews): 1. Observational fieldwork conducted to observe everyday routine activities related to Telehomecare.
  2. In-depth interview conducted for 30-60 min using semi-structured interview guide to assess technician experience with Telehomecare program.

SUMMARY:
The goal of this study is to evaluate the overall impact of Telehomecare on COPD and HF patients and system level outcomes using a comparison group of patients that did not participate in the program (for up to 18 months). This evaluation study will explore costs, participants' experiences, perceptions, and patterns of use related to Telehomecare. The study will include eight Local Health Integration Networks (LHINs) across Ontario, Canada.

DETAILED DESCRIPTION:
The key question to answer is how different models of Telehomecare enabled self-management impacts patient outcomes, experiences and system costs across Ontario. The evaluation study will also attempt to answer questions on who is benefitting the most from the program and the quantifiable benefits a patient would experience from participating.

The intervention evaluation study will use a mixed-methods design comprising of four components (sub-studies), using both qualitative and quantitative research methods: (1) Comparative Effectiveness Study that evaluates patient-level clinical outcomes (e.g. hospitalization, ED visits) using administrative data in comparison with usual care; (2) Economic Evaluation Study that will evaluate costs associated with the program and patient level outcomes as well as cost-effectiveness of the program in comparison with 'usual care'; (3) Evaluation study of Telehomecare use that will evaluate the patterns of program use and perceived quality of life, disease management, satisfaction and caregiver strain; and (4) Adoption study that will use ethnographic fieldwork, semi-structured interviews (during and after program participation) and review of documentary sources to gain understanding of program adoption.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* The patient has a documented diagnosis of HF or COPD (with or without co-morbid conditions);
* The patient has been classified as a 'heavy user' of the health care system, characterized by any of the following:

  * A minimum of one hospitalization for a respiratory or cardiac complaint in the past six months;
  * A minimum of two emergency department/urgent care center visits for a respiratory or cardiac complaint in the past six months;
  * Currently receiving nursing services via CCAC;
  * Frequent visits to primary care provider in the past year;
* Patient/informal caregiver (if applicable) is an adult (over 18 years), able and willing to provide informed consent;
* Patient/informal caregiver (if applicable) is fluent in English;
* Patient/informal caregiver is able and willing to operate the Telehomecare equipment; and
* Patient lives in a residential (private home or retirement home) setting with an active landline.

In addition to the program eligibility criteria, the following criteria for the intervention evaluation study apply to recruitment of patients:

* Patient must have a documented consent for participating in Telehomecare
* Patients enrolled in the Telehomecare program must have agreed to share their contact and health information for evaluative purposes
* Patients must provide informed consent before participating in observations, interviews, and surveys as part of the program evaluation study

Healthcare Provider

A healthcare provider that has:

* Referred a patient that has been previously enrolled in the Telehomecare program, and/or;
* Provided primary care to a patient enrolled in the evaluation study
* Previously or currently participated in delivering Telehomecare as a provider or care administrator; o For observations, interviews, and surveys: nurses/physicians must have at least 2 months experience in providing care using Telehomecare

Technicians, Administrators, and/or Decision Makers

The following are eligible for inclusion in the study:

* Technicians involved in the set-up of Telehomecare equipment in the patient home.
* Administrators and/or decision makers of the Telehomecare program as a larger network of care such as Healthcare Program Managers, key members of the LHINs, OTN etc.

Exclusion Criteria:

Patient

* Less than 18 years of age;
* Individuals without an established diagnosis of COPD or HF
* Unable or unwilling to provide verbal informed consent
* Demonstrated non-adherence to the THC program:

  o The Telehomecare Nurse works with each patient on a case-by-case review to assess willingness to partner in their own care, and if the number of missed consultation appointments and reasons for demonstrate overall non-adherence with the program;
* Inability or unwillingness to use Telehomecare equipment, and/or;
* Do not have a regular caregiver to assist in the use of the equipment (if assistance is required)

Healthcare Provider

* Is not a practicing healthcare provider in any of the said LHINs

Technicians, Administrators and/or Decision Makers

* Unable or unwilling to provide verbal informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This community based study will be conducted across 8 Local Health Integration Networks (LHINs) in Ontario: Toronto Central, North East, Central West, Erie St Claire, Central, North Simcoe Muskoka, North West and South West LHINs.
  The study population will include COPD and HF patients that currently or previously participated in Telehomecare program. The study population will also include informal caregivers and healthcare providers involved in and/or caring for a patient enrolled in the program as well as administrators /decision makers involved with the Telehomecare program.
Sampling Method: Probability Sample
Enrollment: 5400 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Disease specific hospitalization and ED visits | 18 months
  Comparison of disease specific hospitalization and ED visits between patients receiving Telehomecare vs. 'usual care' (followed up to 18 months)

SECONDARY OUTCOMES:
Number of all-cause hospitalization/ED visits | 18 months
  Comparison of the number of all-cause hospitalization/ED visits between patients receiving Telehomecare vs. 'usual care' (followed up to 18 months)
Number of visits to primary care physicians | 18 months
  Comparison of the number of visits to primary care physicians between patients receiving Telehomecare vs. 'usual care' (followed up to 18 months)
Number of visits to specialists | 18 months
  Comparison of the number of visits to specialists between patients receiving Telehomecare vs. 'usual care' (followed up to 18 months)
Number of visits to in-home health professionals | 18 months
  Comparison of the number of visits to in-home health professionals between patients receiving Telehomecare vs. 'usual care' (followed up to 18 months)
Number of admissions to long-term care facilities | 18 months
  Comparison of the number of admissions to long-term care facilities between patients receiving Telehomecare vs. 'usual care' (followed up to 18 months)
Length of stay in hospital | 18 months
  Comparison of length-of-stay in hospital between patients receiving Telehomecare vs. 'usual care' (followed up to 18 months)
Medication use | 18 months
  Comparison of medication use between patients receiving Telehomecare vs. 'usual care' (followed up to 18 months)

OTHER OUTCOMES:
Costs associated with Telehomecare equipment and services | 18 months
  Costs associated with Telehomecare equipment and services; comparison of health services costs for Telehomecare and 'usual care'; incremental cost-effectiveness ratio (ICER) of Telehomecare compared with 'usual care'
Comparison of health services costs for Telehomecare and 'usual care' | 18 months
  Costs associated with Telehomecare equipment and services; comparison of health services costs for Telehomecare and 'usual care'; incremental cost-effectiveness ratio (ICER) of Telehomecare compared with 'usual care'
Incremental cost-effectiveness ratio (ICER) of Telehomecare compared with 'usual care' | 18 months
  Costs associated with Telehomecare equipment and services; comparison of health services costs for Telehomecare and 'usual care'; incremental cost-effectiveness ratio (ICER) of Telehomecare compared with 'usual care'
Patterns of use of the program | 12 months
  Patterns of use of the program; patient quality of life, disease self-management skills and satisfaction with Telehomecare; Informal caregivers strain
Patient quality of life, disease self-management skills and satisfaction with Telehomecare | 12 months
  Patterns of use of the program; patient quality of life, disease self-management skills and satisfaction with Telehomecare; Informal caregivers strain
Informal caregivers strain | 12 months
  Patterns of use of the program; patient quality of life, disease self-management skills and satisfaction with Telehomecare; Informal caregivers strain
Perceptions and experiences of patients | 12 months
  Perceptions and experiences of patients, informal caregivers, providers, administrators/decision-makers; overall adoption, integration and sustainability of the program
Overall adoption, integration and sustainability of the program | 12 months
  Perceptions and experiences of patients, informal caregivers, providers, administrators/decision-makers; overall adoption, integration and sustainability of the program

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Rac, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No